CLINICAL TRIAL: NCT06420206
Title: Goals of Care Discussion for Patients With Advanced Lung and Gastrointestinal Cancer in the Emergency Department of a Comprehensive Cancer Center
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-1024
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Lung Neoplasms; Gastrointestinal Neoplasms | interventions — Standard of Care; Patient Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Cancer Care Center (Other): In Group 1, participants will receive the usual standard of care, during your emergency room visit, provided by the Acute Cancer Care Center (ACCC) treating doctor who will address symptoms and other medical problems that brought the participant to the emergency room.
  Interventions: Other: Standard of Care (Acute Cancer Care Center)
- Goals of Care (Other): In Group 2, participants will receive the above usual standard of care plus goals of care (GOC) intervention.
  Interventions: Other: Standard of Care (Goals of Care)

INTERVENTIONS:
Other: Standard of Care (Acute Cancer Care Center) — In Group 1, participants will receive the usual standard of care by an emergency care physician not trained in palliative care.
  Arms: Acute Cancer Care Center
Other: Standard of Care (Goals of Care) — In Group 2, participants will receive standard of care plus palliative care intervention by an emergency care physician trained in palliative care.
  Arms: Goals of Care

SUMMARY:
To improve quality of life for participants with advanced cancer, support their families, and lower overall cost of care.

DETAILED DESCRIPTION:
Primary Objective:

To compare overall percentage of days spent in an acute care setting over the 30-day period from time of the index emergency department (ED), referred to as Acute Cancer Care Center (ACCC), visit for patients who receive the emergency department-based GOC intervention and those who do not.

Secondary Objective:

To obtain data on rates of admission to the ICU, death in the hospital setting, symptom improvement for participants hospitalized, hospice referral, survival, and 30-day care costs for participants who receive the GOC intervention in the ACCC and those who do not.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is at least 18 years old presenting to the triage area of the MDACC ACCC for treatment
2. Participant has advanced lung or GI cancer. Advanced cancer patient defined as: locally recurrent or metastatic for which there is no curative treatment available.
3. Participant screens positive for at least 2 of 3 triple threat conditions (dyspnea, altered mental status, or poor performance status)
4. Participant has the ability to speak and write in English
5. Participant has the ability to provide consent OR is accompanied by a LAR able to provide consent

Exclusion Criteria:

1. Participant is already enrolled in hospice
2. Participant is comatose
3. Participant has severe intellectual disability
4. Participant has a history of dementia documented in the medical records
5. Participant has baseline communication barriers such as aphasia or deafness
6. Participant is new to MDACC, without established oncology care at our institution at time of ACCC arrival
7. Participant is 18 years or older, currently cared for by pediatrics service
8. Pregnant women
9. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Quality Of Life Questionnaire | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elsayem, MD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org